CLINICAL TRIAL: NCT04324931
Title: Effect of Biomechanical Corrections of Tibia on Medial Joint Space Loading, Varus Deformity and Functional Tasks in Patients With Medial Tibiofemoral Joint Osteoarthritis: A Quasi-Experimental Study
Brief Title: Effect of Biomechanical Correction in Medial Tibiofemoral Joint Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate Professor Maharishi Markandeshwar (Deemed to be university), Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMDU/IEC/1527; U1111-1249-3661 (Other: World Health Organization)
Record Dates: First submitted 2020-03-06; First posted 2020-03-27 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis Knee
Keywords: Obesity; Osteoarthritis; Physical Therapy Modalities
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Single Group pre-test, post-test design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biomechanical corrections (Experimental): In this group, biomechanical correction will be perform with the help of mobilization with movement to correct biomechanical misalignment and along with this conventional treatment, in which Hydrocollatoral packs for 20 minutes, Interferential Therapy for 15 minutes with beat frequency 100 Hz, Sweep frequency 150 Hz and exercise program for 3 sessions of 20 minutes on alternative days for 3 weeks. Which will be given for three days a week for three weeks.
  Interventions: Other: Biomechanical corrections; Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Biomechanical corrections — Biomechanical corrections is to be done to correct the varus deformity of knee joint and for pain management.
Other: Conventional Physiotherapy — Conventional therapy includes Hydrocollatoral pack for 20 minutes, Interferential therapy for 15 minutes beat frequency 100 Hz, Sweep frequency 150 Hz and exercise program of 3 sessions for 20 minutes on alternative days for 3 weeks for management of knee osteoarthritis.

SUMMARY:
Effect of Biomechanical Correction of Tibia on Medial Joint space loading, Varus deformity and functional tasks in patients with medial tibiofemoral joint osteoarthritis in which participants will be taken. The outcome measures taken are Trauma CAD Software, NPRS, WOMAC and Goniometery will be measured at the baseline after 3rd week of the intervention.

DETAILED DESCRIPTION:
Background: Knee osteoarthritis (KOA) are very prevalent chronic disease of the joint which causing the functional disability and pain specifically in older adults.

Objective: Purpose of the study is to see that the biomechanical correction on the tibia and varus deformity is effective in the conventional treatment of participants with the KOA.

Study Design: A Randomized single group Pretest-Post test Clinical Trial. Methodology: Total '5' subjects were included in the study with the age of 40 to 60 years based on exclusion and inclusion criteria. For the pain, the NPRS will be taken, goniometer taken for the measurement of range of motion, WOMAC will be taken for the physical activity measurement and CAD Software will be taken to see the alignment of the affected limb. Conventional treatment will also be given.

Conclusion: Biomechanical correction shows the significant improvement and improves the subject's physical activity and reduces the pain and stiffness.

Keywords: Obesity, Osteoarthritis, Pain and Physical therapy modalities

ELIGIBILITY:
Inclusion Criteria: • 40-60 years of age paients will be included in this study

* BMI (25.1±4.2) kg/m2
* Subjects with stiffness and knee pain
* Subjects with objection of pain in knee joint that was aggravated by performing 2 or more of the following functional activities: prolonged cross sitting, stair assents and descent, squatting and kneeling.
* Subjects who are willing to take participation
* Individuals who obeys the commands properly
* Individuals exhibiting the subsequent biomechanical changes on screening
* Q angle >12 degree for male and >15 degree for female, femoral anteversion, external tibial torsion >15 degree, lack of ≥ 5 degree of knee extension in supine position.

Exclusion Criteria:

* • Knee meniscal injuries or ligament injuries

  * Lately history of lower limb trauma and surgery
  * In recent times fracture in lower extremity
  * In lower extremity metal plantation
  * Cardio vascular conditions
  * Patella Dislocation/subluxation
  * Abnormality in foot or deformity

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in lower limb alignment by Trauma CAD software | Baseline, 3 weeks after intervention
  Trauma CAD Software will be used to measure the misalignment of the lower limb

SECONDARY OUTCOMES:
Change in pain level by Numeric Pain Rating Scale | Baseline, 3 weeks after intervention
  This scale will be used for assessment of pain
Change in joint range of motion by Goniometery | Baseline, 3 weeks after intervention
  Use for range of motion measurement
Change in physical performance | Baseline, 3 weeks after intervention
  WOMAC will be used for assessment

CONTACTS AND LOCATIONS:
Overall Officials: Sunaina Saini, BPT, Principal Investigator — Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation
Locations (1):
- Sunaina Saini, Kurukshetra, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pal CP, Singh P, Chaturvedi S, Pruthi KK, Vij A. Epidemiology of knee osteoarthritis in India and related factors. Indian J Orthop. 2016 Sep;50(5):518-522. doi: 10.4103/0019-5413.189608. PMID 27746495
- [Result] Crema MD, Felson DT, Guermazi A, Nevitt MC, Niu J, Lynch JA, Marra MD, Torner J, Lewis CE, Roemer FW. Is the atrophic phenotype of tibiofemoral osteoarthritis associated with faster progression of disease? The MOST study. Osteoarthritis Cartilage. 2017 Oct;25(10):1647-1653. doi: 10.1016/j.joca.2017.05.019. Epub 2017 Jun 9. PMID 28606556
- [Result] Felson DT, Goggins J, Niu J, Zhang Y, Hunter DJ. The effect of body weight on progression of knee osteoarthritis is dependent on alignment. Arthritis Rheum. 2004 Dec;50(12):3904-9. doi: 10.1002/art.20726. PMID 15593215
- See also: This study has evidenced a large percentage of population as borderline OA; therefore, it depends mainly on the prevention of modifiable risk factors to preserve at ease movement in elderly population through awareness programs. — https://www.ncbi.nlm.nih.gov/pubmed/27746495
- See also: the atrophic phenotype of knee OA was associated with a decreased likelihood of progression of JSN and cartilage loss compared to the non-atrophic knee OA phenotype. — https://www.ncbi.nlm.nih.gov/pubmed/28606556
- See also: Although elevated BMI increases the risk of knee OA progression, the effect of BMI is limited to knees in which moderate malalignment exists, presumably because of the combined focus of load from malalignment and the excess load from increased weight. — https://www.ncbi.nlm.nih.gov/pubmed/15593215